CLINICAL TRIAL: NCT02279836
Title: Open Label, Multi-center, Single Arm Post-marketing Study of SC20 Colonoscope and Colonoscopy System for Colonoscopy in Male and Female Patients >18 Years Old
Brief Title: Single Arm Post-marketing Study of SC20 Colonoscope
Acronym: SC20 Scope
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped due to the expected introduction of a next product generation.
Sponsor: Invendo Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Invendo s14-01040
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Gentle Colonoscopy
Keywords: Patients with any indication for colonoscopy in the U.S.A.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm post-marketing Study (Other): SC20 Colonoscope and Colonoscopy System For Colonoscopy
  Interventions: Device: SC20 Colonoscope

INTERVENTIONS:
Device: SC20 Colonoscope — Single Arm Post-Marketing Study of SC20 Colonoscope

SUMMARY:
The objective of the study is to gather post-market data regarding the performance of the invendo SC20 colonoscope in a real-world US population.

DETAILED DESCRIPTION:
The objective of the study is to expand data collection and product exposure in a controlled clinical setting and gather data regarding the performance of the Invendo SC20 colonoscope in a real-world US population. The objective of the study is to specifically monitor three points:

1. The diagnostic performance of the device including polyp and adenoma detection rates;
2. The therapeutic performance of the device (the ability of the physician to remove/biopsy identified lesions);
3. Performance of the device in a typical colonoscopy population, including patients with underlying inflammatory bowel disease (IBD), previous pelvic surgery or irradiation, obesity, diverticular disease, and previous colorectal surgery, as they present in the study population (see below C.).

ELIGIBILITY:
Inclusion Criteria:

* Any indication for colonoscopy
* Willing to give informed consent
* Willing to consume 2-4 liters of bowel prep

Exclusion Criteria:

* An age younger than 18 years
* Congestive heart failure
* Renal insufficiency
* Intestinal obstruction
* Any acute life-threatening condition (in the opinion of the investigator)
* Current pregnancy
* Abdominal surgery in the past 6 months
* Bleeding disorders
* Inability to provide informed consent
* Any other contraindication to colonoscopy (e.g. fulminant colitis or acute diverticulitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
1. Cecal intubation rates (visualization of the cecum by notation of landmarks and photo documentation of landmarks in every procedure) | average 6 to 12 months

SECONDARY OUTCOMES:
2. Detection of polyps, adenomas and other lesions in all individuals | average 6 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Goodman, MD, Principal Investigator — NYU Langone Medical Center
Locations (3):
- United States (3):
  - Bellevue Hospital Center, New York, New York
  - NYU Langone Medical Center Ambulatory care, New York, New York
  - New York Presbyterian Columbia University Medical Center, New York, New York